CLINICAL TRIAL: NCT04554862
Title: The Analgesic Efficacy of Adding Magnesium Sulfate Versus Ketorolac to Bupivacaine in Ultrasound-guided Supraclavicular Brachial Plexus Block (A Prospective- Double-blinded Randomized Controlled Trial)
Brief Title: The Analgesic Efficacy of Magnesium and Ketorolac in Ultrasound Supraclavicular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Safaa Gaber Ragab, Lecturer of anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M419
Record Dates: First submitted 2020-09-13; First posted 2020-09-18 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
Keywords: Magnesium; Ketorolac; Supraclavicular block
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (M) magnesium sulfate (Active Comparator): a 6ml of magnesium sulfate 10% (600mg) will be added to 25ml of bupivacaine 0.5% for supraclavicular brachial plexus block
  Interventions: Drug: Magnesium sulfate; Procedure: supraclavicular block
- the intervention group (K) ketorolac (Active Comparator): a 2ml of ketorolac (30mg) will be added to 4ml of normal saline and 25ml of bupivacaine 0.5% for supraclavicular brachial plexus block
  Interventions: Drug: Ketorolac Tromethamine; Procedure: supraclavicular block

INTERVENTIONS:
Drug: Magnesium sulfate — magnesium sulfate will be added to the block
  Other Names: magnesium 10%
  Arms: the intervention group (M) magnesium sulfate
Drug: Ketorolac Tromethamine — ketorolac will be added to the block
  Other Names: ketorolac
  Arms: the intervention group (K) ketorolac
Procedure: supraclavicular block — it is done by ultrasound- guided

SUMMARY:
Despite many regional anesthetic techniques have been described for anesthesia of the brachial plexus which is responsible for the sensory and motor innervation of entire upper limb, still, supraclavicular block (SCB) is the regional anesthetic technique of choice.

SCB has been described as the spinal anesthesia of the upper limb as it offers dense anesthesia of the brachial plexus for the surgical procedures below the arm from elbow to hand. Although the SCB has a high incidence of complications like pneumothorax, the use of ultrasound-guided block improved the safety for the patient. There are several adjuvants have been added to SCB aiming for prolongation of the duration of peripheral nerve block as fentanyl, alpha 2 adrenergic agonist (Dexmedetomidine, Clonidine), tramadol, ketorolac and Magnesium sulfate.

Magnesium has anti-nociceptive effects in animal and human models, principally related to blocking the N-methyl-D-aspartate (NMDA) receptors and regulation of calcium influx into cells. Calcium influx leads to a sequence of central sensitization such as windup phenomenon and long term potentiation which are crucial mechanisms that determine the duration and intensity of post-operative pain. Magnesium prevents central sensitization triggered by peripheral nociceptive stimulation in response to painful stimuli.

Non-Steroidal Anti-Inflammatory drugs (NSAID) inhibit synthesis of prostaglandins from arachnoid acid in phospholipid membranes resulting in decreased afferent nociceptive signals from the site of surgery. There are a lot of studies supported the analgesic effect when NSAIDs are concentrated at a peripheral site compared to the systemic administration therapy. Ketorolac is a parenteral NSAIDs. Studies have shown that ketorolac as an adjuvant to local anesthetics during peripheral nerve block enhanced duration and quality of analgesia.

DETAILED DESCRIPTION:
Eighty adult patients scheduled for upper limb surgeries from elbow to hand will be enrolled in the study after obtaining approval of the local institutional ethics committee and local institutional review board at Fayoum University Hospital. A detailed informed consent will be signed by the eligible participants before recruitment and randomization.

80 patients will be chosen to receive either Mg (group M, n=40) or ketorolac (group K, n=40) randomly by a computer-generated table. The randomization sequence will be concealed in opaque sealed envelopes. The envelopes will be opened by the study investigator just after recruitments and admission to the operation room. Only participants and care providers will be blinded to the group allocations. The consolidated standards of reporting trials (CONSORT) recommendations for reporting randomized, controlled clinical trials will be followed.

Patient preoperative preparations:

Preoperative investigations will be done according to the local protocol designed to evaluate the patients. It will include complete blood count, blood sugar level, serum urea and creatinine, liver function tests, coagulation profile, and ECG.

Before surgery, the participants will receive education about the (NRS) from (0-10 mm) (where 0=no pain and 10 = worst comprehensible pain) and the details of the nerve block procedures.

After a 6h fasting, the patients will be taken to the operating theatre.

Anesthetic technique:

A (20G) IV catheter will be placed in the UL opposite the surgical site after the arrival of the patient to the operating room. IV premedication will be administered to all patients (midazolam 0.02mg/kg and fentanyl 50mcg/dose). Supplemental oxygen (nasal cannula at 2L/min), and standard ASA monitoring (5-lead ECG, NIBP, and pulse oximetry) will be applied throughout the procedure.

Block technique

For the ultrasound-guided SCB, the patients will be placed in a supine position and the head turned slightly to the opposite side of their block. The injured hand will be put on the patient's abdomen and the shoulder will be moved downward as much as possible. The supraclavicular area will be cleaned using an antiseptic iodine solution and draped. Once the skin will be appropriately cleaned and prepared with anti-septic, the high-frequency linear array transducer will be placed over the supraclavicular area. After infiltration of the site by a local anesthetic, a sterile 22 gauge, 50 mm echogenic needle under ultrasound guidance will be inserted and after reaching the tip of the needle near the subclavian artery around the brachial plexus, the solution will be injected and the spread of the drug will be visualized. 25 ml of bupivacaine 0.5% + 6ml of magnesium sulfate 10% will be injected to group M and 25ml of bupivacaine 0.5% + 2ml of ketorolac 30mg + 4ml normal saline will injected to group K. The continuous aspiration and injection will be taken to avoid intravascular injection. After performing the block on the patients, hemodynamic parameters and all complications related to SCB (pneumothorax, hematoma, hypotension, bradycardia, etc.) will be recorded. After ensuring adequate anesthetic effect of the block, the surgery was started.

Assessment of sensory and motor blockade:

The extent of motor and sensory blockade will be evaluated by an anesthesiologist who will not be involved in the SCB 30 minutes. after local anesthetic administration. Using an alcohol swab, the sensory blockade will be tested by pin prick test using a 3- point scale:

Grade 0: normal sensation. Grade 1: decreased pain sensation to pinprick. Grade 2: loss of pain sensation to pinprick in the median, ulnar, radial and musculocutaneous nerve locations.

And it will be tested every 5 minutes for 30 minutes.

Motor blockade will be assessed by using (modified bromage) 3-point scale:

Grade 0: Normal motor function. Grade 1: Decreased motor strength with ability to move fingers only. Grade 2: Complete motor block. And it will be tested every 5 minutes for 30 minutes. When the operation was over, NRS score will be measured at 0, 1, 4, 8, 12, 24 hours.

Post-operative care:

Patients will be transferred to post-anesthetic care unit (PACU) for 2 hours. Then the patients will be discharged from the PACU.

Patient will receive analgesic according to the local institutional protocol as the following (Diclofenac sodium 75mg and paracetamol 1 gram by intravenous infusion over 30 minute.) as a component of multimodal anesthesia regimen for postoperative pain control.

Post-operative pain will be rated on (NRS) from 0 (no pain) to 10 (worst imaginable pain) at 1hr at PACU then at 4,8,12 and 24 hours postoperatively.

Patients with NRS>5 will receive morphine sulfate IV at a bolus dose of 2-5 mg increments with maximum dose of 20 mg at 4hours or 40mg at 24 hours. The morphine titration protocol will be suspended with Oxygen saturation < 95%; Respiratory rate < 10 / minute; the development of sedation (Ramsay sedation scale >2); development of acute adverse effects (allergy, marked itching, excessive vomiting, and hypotension with systolic blood pressure less than 20% of baseline values); or attaining adequate level of analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status from I to III participants who were scheduled for surgical procedures of the arm from elbow to hand

Exclusion Criteria:

* Patient refusal.
* Contraindication to regional anesthesia (coagulopathy, allergy to the local anesthetic or any adjuvants added, severe thrombocytopenia, pre-existing neuropathy in the operative limb, infection at puncture site).
* Sepsis.
* Pregnant or lactating women.
* Hepatic or renal dysfunction.
* Any drug or opioid abuse.
* Surgical procedures for more than 3h.
* Advanced cardiac diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
the cumulative morphine consumption | At 24 hours postoperative
  In milligrams

SECONDARY OUTCOMES:
numerical rating scale (NRS) of postoperative pain | at 1 hour in the post-anesthesia care unit (PACU)
  the severity of postoperative pain estimated by numerical rating scale (NRS) ( where 0 = no pain and 10 = worst imaginable pain)
numerical rating scale (NRS) of postoperative pain | at 4 hours postoperative
  the severity of postoperative pain estimated by numerical rating scale (NRS) ( where 0 = no pain and 10 = worst imaginable pain)
numerical rating scale (NRS) of postoperative pain | at 8 hours postoperative
  the severity of postoperative pain estimated by numerical rating scale (NRS) ( where 0 = no pain and 10 = worst imaginable pain)
numerical rating scale (NRS) of postoperative pain | at 12 hours postoperative
  the severity of postoperative pain estimated by numerical rating scale (NRS) ( where 0 = no pain and 10 = worst imaginable pain)
numerical rating scale (NRS) of postoperative pain | at 24 hours postoperative
  the severity of postoperative pain estimated by numerical rating scale (NRS) ( where 0 = no pain and 10 = worst imaginable pain)
incidence of opioid related side-effects | 5 minutes after supraclavicular block till discharge from PACU
  side effects (nausea, vomiting, pruritus, excessive sedation, and respiratory depression)
incidence of adverse effects related to the block | 5 minutes after supraclavicular block till discharge from PACU
  adverse events (e.g. vascular puncture, local anesthetic toxicity, and pneumothorax)
time to the first requirement of analgesic supplement | 5 minutes After supraclavicular block till first requirement of analgesic
  In minutes
Duration of surgical procedures | 5 minutes after completion of surgical procedures
  In minutes
Assessment of heart rate | from the start of the block till completion of surgical procedures
  In beats per minutes
Assessment of mean blood pressure | from the start of the block till completion of surgical procedures
  In millimetre mercury (mmHg)
Assessment of respiratory rate | from the start of the block till completion of surgical procedures
  Number of breaths per minute
Assessment of Oxygen saturation | from the start of the block till completion of surgical procedures
  In percentage through use of pulse oximetry
Age | 10 minutes before surgery
  in years
Weight | 10 minutes before surgery
  in kilograms (kg)
Height | 10 minutes before surgery
  in meters (m)
Body mass index | 10 minutes before surgery
  in kg/m square

CONTACTS AND LOCATIONS:
Overall Officials: Safaa G Ragab, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

REFERENCES:
- [Background] Mukherjee K, Das A, Basunia SR, Dutta S, Mandal P, Mukherjee A. Evaluation of Magnesium as an adjuvant in Ropivacaine-induced supraclavicular brachial plexus block: A prospective, double-blinded randomized controlled study. J Res Pharm Pract. 2014 Oct;3(4):123-9. doi: 10.4103/2279-042X.145387. PMID 25535620
- [Background] Mirkheshti A, Saadatniaki A, Salimi A, Manafi Rasi A, Memary E, Yahyaei H. Effects of dexmedetomidine versus ketorolac as local anesthetic adjuvants on the onset and duration of infraclavicular brachial plexus block. Anesth Pain Med. 2014 Aug 2;4(3):e17620. doi: 10.5812/aapm.17620. eCollection 2014 Aug. PMID 25237638
- [Background] Lee AR, Yi HW, Chung IS, Ko JS, Ahn HJ, Gwak MS, Choi DH, Choi SJ. Magnesium added to bupivacaine prolongs the duration of analgesia after interscalene nerve block. Can J Anaesth. 2012 Jan;59(1):21-7. doi: 10.1007/s12630-011-9604-5. Epub 2011 Oct 20. PMID 22012543
- [Background] Reinhart DJ, Stagg KS, Walker KG, Wang WP, Parker CM, Jackson HH, Walker EB. Postoperative analgesia after peripheral nerve block for podiatric surgery: clinical efficacy and chemical stability of lidocaine alone versus lidocaine plus ketorolac. Reg Anesth Pain Med. 2000 Sep-Oct;25(5):506-13. doi: 10.1053/rapm.2000.7624. PMID 11009237
- [Background] Akhondzade R, Nesioonpour S, Gousheh M, Soltani F, Davarimoghadam M. The Effect of Magnesium Sulfate on Postoperative Pain in Upper Limb Surgeries by Supraclavicular Block Under Ultrasound Guidance. Anesth Pain Med. 2017 Jun 10;7(3):e14232. doi: 10.5812/aapm.14232. eCollection 2017 Jun. PMID 28924560